CLINICAL TRIAL: NCT05502900
Title: Adjuvant Melatonin for Uveal Melanoma: A Randomized Open Phase III Study
Brief Title: Adjuvant Melatonin for Uveal Melanoma
Acronym: AMUM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustav Stalhammar (Other)
Collaborators: Karolinska Trial Alliance (Industry); The Swedish Eye Foundation (Ögonfonden) (Unknown); The Swedish Society of Medicine (Other); Swedish Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Gustav Stalhammar, M.D. Ph.D., St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMUM v 2.0; 2022-500307-49 (EudraCT Number)
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Uveal Melanoma; Uveal Melanoma, Posterior, Medium/Large Size; Eye Cancer, Intraocular Melanoma
Keywords: Melatonin; Adjuvant; Preventive; Uveal melanoma; Survival; Phase 3 trial
MeSH Terms: conditions — Uveal Melanoma | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: 100 patients will be randomized into either adjuvant treatment with Melatonin or to a control group that will undergo standard follow-up with radiological examinations but no adjuvant treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Experimental): Melatonin tablet 5 mg. 4 tablets taken at night (20 mg) for 5 years.
  Interventions: Drug: Melatonin
- Control (No Intervention): No intervention. Follows the current standard of observation after primary tumor treatment.

INTERVENTIONS:
Drug: Melatonin — White round tablets, each with a dose of 5 mg Melatonin. 4 tablets taken simultaneously at night. Tablets can be crushed and/or taken with a glass of water if the patient wish.
  Other Names: Melatonin AGB Pharma
  Arms: Melatonin

SUMMARY:
Uveal melanoma (UM) is the most common type of cancer inside the eyes of adults. Almost half of all patients diagnosed with UM will eventually develop metastases. Once metastases occur, the median patient survival is short.

In this trial, we will test if treatment with Melatonin after primary tumor diagnosis can prevent or delay the development of metastases. 100 patients diagnosed with primary UM will be randomized to either treatment with Melatonin tablets (20 mg at night), or to a control group. Both groups will be followed for 5 years. At 5 years, the number of patients that have developed metastases in the Melatonin and control groups will be compared (primary outcome measure).

DETAILED DESCRIPTION:
At the time of primary UM diagnosis, about 2 % of patients have radiologically detectable metastases. Within 15 years, this proportion increases to 32-45 % even with successful treatment of the eye. Presumably, this is caused by subclinical dormant micrometastases that most frequently locate to the liver. Once these leave their dormant state and grow into clinically detectable lesions, few effective treatment alternatives are available and the median patient survival is about one year.

Several trials have tested interventions for metastatic UM, and in comparison with the greatly improved results for cutaneous melanoma during the last decades, response rates and durations have been low.

The AMUM trial will therefore test if adjuvant treatment with Melatonin for 5 years after primary tumor diagnosis can prevent or delay the onset of metastases. 100 patients recently diagnosed with primary UM and found to have a high risk of metastasis will be recruited. The trial is administered from St. Erik Eye Hospital, Stockholm, Sweden, who has a national responsibility for the diagnosis, plaque brachytherapy treatment and histopathological examination of uveal melanomas. This means that all Swedish patients that are diagnosed with uveal melanoma may be considered for inclusion in the trial, regardless of their region of residence. Patients will be screened for eligibility, informed, recruited, randomized, and treated from St. Erik Eye Hospital. Follow-up will be conducted in cooperation with multiple centers all over the country.

When informed consent has been obtained, the 100 patients will then be randomized to either treatment with oral tablets of Melatonin (20 mg, taken before bedtime) for 5 years, or to a control group. Both groups will be followed with regular contacts from the investigators, with radiological examinations of the liver every 6 months, and with a blood test at the time of recruitment and then year 2 and 4.

When the last patient has taken his or her last tablet after 5 years of treatment, we will examine the primary outcome measure (relative risk of metastasis) and secondary outcome measures (overall survival, survival after development of metastases, number of patients developing other cancers, adverse events (AE) and serious adverse events (SAE)) in the Melatonin vs. control arm.

AMUM is an Investigator-Initiated Trial without commercial interests.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥18 years
2. The patient has given his/her written informed consent to participate in the trial.
3. The patient has a melanoma originating in the choroid or in the ciliary body, as diagnosed by clinical methods and/or histological examination.

   AND at least one of the following 7 items:
4. The patient's tumor is of size category T3d or higher, or stage IIIB or IIIC according to the American Joint Committee on Cancer (AJCC, version 8) criteria.
5. The patient's tumor is large according to modified criteria from the Collaborative Ocular Melanoma Study (COMS), i.e. largest basal diameter >16 mm or apical thickness >8 mm.
6. The patient's tumor was of size category T2a before plaque brachytherapy and has then recurred.
7. The patient's tumor has an epithelioid cell type (>5 epithelioid cells per high power field and >90 % of tumor cells epithelioid).
8. The patient's tumor has a low immunohistochemical expression of BAP1.
9. The patient's tumor has more than 9 mitoses per high power field.
10. The patient has >60 % risk of metastases within 5 years, as determined with another published and validated prognostic test (e.g. gene expression class 2).
11. If the patient is already being treated with Melatonin, a two-week wash out period will be applied before randomization.

Exclusion Criteria:

1. Oversensitivity or allergy to Melatonin or any of the excipients in the tablet.
2. The patient has metastatic disease, detectable with radiological examinations or any other method (development of metastases after recruitment to the trial does not disqualify the patient from participation).
3. The patient is unable to provide informed consent.
4. The patient has decreased liver function (e.g., liver cirrhosis or hepatitis)
5. The patient is pregnant or a fertile woman (Women of child-bearing potential, WOCBP). Fertility is defined as the time between menarche and menopause for women that are not permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy. Menopause is defined as absence of menstruation for 12 months or longer without other cause.
6. The patient is breast feeding or is planning to breastfeed before the end of the trial. Women that are included in the trial and begin to breastfeed before the end of the trial must resign from the trial.
7. The patient has epilepsy.
8. The patient is being treated (for more than 4 weeks) with CYP1A2 inhibitors Fluvoxamine, Ciprofloxacin, Norfloxacin, or Verapamil, with combined hormonal contraception (containing etinylestradiole and progestin), with hormonal substitution therapy, with 5- or 8-metoxypsoralene or cimetidine. If a patient starts using any of these substances for more than 4 weeks after recruitment to the trial, he or she does not need to resign from the trial but may pause the use of Melatonin, and then restart after the use of the other substance has ceased. Concurrent treatment with CYP1A2 inducers including carbamazepine, fenytoine, rifampicin, omeprazole, calcium antagonists, benzodiazepine-related hypnotics, non-steroid anti-inflammatory drugs (NSAIDs) and beta blockers is not an exclusion criterium. Concurrent treatment with warfarin or other vitamin K antagonists is not an exclusion criterium, but requires information to the patient and discussion about dose adjustments with the prescribing physician.
9. The primary UM was diagnosed more than 12 months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-02 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that develop metastases in Melatonin vs. Control arm, evaluated as relative risk (RR). | 5 years
  Measured as relative risk (i.e., the incidence rate of metastasis in the Melatonin arm divided by the incidence rate in the control group), with 95 % confidence interval.

SECONDARY OUTCOMES:
Number of patients that develop metastases in Melatonin vs. Control arm, evaluated as Cox regression hazard ratio (HR). | 5 years
  Measured as hazard ratio (i.e., the hazard for metastasis in the Melatonin arm divided by the hazard in the control group) with relevant covariates (e.g., tumor size, patient age, BAP-1 expression), with 95 % confidence interval.
Overall survival (OS) time from randomization in Melatonin vs. Control arm, evaluated with the Log-rank test. | 5 years
  Overall survival (the length of time from randomization that patients are still alive) in the Melatonin vs. Control arm. A Kaplan-Meier-curve will be drawn and the Log-rank test will be applied.
Overall survival (OS) time from the detection of metastasis in Melatonin vs. Control arm, evaluated with the Log-rank test. | 5 years
  Overall survival (the length of time from radiological detection of metastases that patients are still alive) in the Melatonin vs. Control arm. A Kaplan-Meier-curve will be drawn and the Log-rank test will be applied.
Number of patients that develop other cancers (i.e., cancer diagnoses other than uveal melanoma) in Melatonin vs. Control arm, evaluated as relative risk (RR). | 5 years
  Measured as relative risk (i.e., the incidence rate of other cancers in the Melatonin arm divided by the incidence rate in the control group), with a 95 % confidence interval.
Number of patients that develop other cancers (i.e., cancer diagnoses other than uveal melanoma) in Melatonin vs. Control arm, evaluated as Cox regression hazard ratio (HR). | 5 years
  Measured as hazard ratio (i.e., the hazard for other cancers in the Melatonin arm divided by the hazard in the control group) with relevant covariates (e.g., tumor size, patient age, BAP-1 expression), with 95 % confidence interval.
Number of participants with treatment-related adverse events (AEs) and serious adverse events (SAEs) in Melatonin vs. Control arm, as assessed by CTCAE v5.0. | 5 years
  Frequency of adverse events (AEs) and serious adverse events (SAEs) in the Melatonin vs. Control arm, evaluated as relative risk (RR) with 95 % confidence interval.

OTHER OUTCOMES:
Interim analysis: Number of patients that develop metastases in Melatonin vs. Control arm, evaluated as relative risk (RR). | 3 years
  Measured as relative risk (i.e., the incidence rate of metastasis in the Melatonin arm divided by the incidence rate in the control group), with 95 % confidence interval.
Interim analysis: Overall survival (OS) in Melatonin vs. Control arm, evaluated with the Log-rank test. | 3 years
  Overall survival in the Melatonin vs. Control arm

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Stålhammar, MD PhD, Principal Investigator — St. Erik Eye Hospital and Karolinska Institutet
Locations (1):
- St. Erik Eye Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kal Omar R, Hagstrom A, Stalhammar G. Adjuvant melatonin for uveal melanoma (AMUM): protocol for a randomized open-label phase III study. Trials. 2023 Mar 26;24(1):230. doi: 10.1186/s13063-023-07245-9. PMID 36966349
- [Background] Hagstrom A, Kal Omar R, Williams PA, Stalhammar G. The rationale for treating uveal melanoma with adjuvant melatonin: a review of the literature. BMC Cancer. 2022 Apr 13;22(1):398. doi: 10.1186/s12885-022-09464-w. PMID 35413810
- See also: Adjuvant melatonin for uveal melanoma (AMUM): protocol for a randomized open-label phase III study — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-023-07245-9